CLINICAL TRIAL: NCT05166486
Title: The Effect of Calisthenic Exercise on Aerobic Capacity, Muscle Strength and Quality of Life in Hemodialysis Patients: a Single-blind Placebo-controlled Randomized Trial
Brief Title: The Effect of Calisthenic Exercise on Aerobic Capacity, Muscle Strength and Quality of Life in Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Nazan Ozturk, Principal Investigator, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Elifibo22
Record Dates: First submitted 2021-11-25; First posted 2021-12-22 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Physical Activity; Patient; Quality of Life; Hemodialysis
Keywords: Exercise; Hemodialysis; Quality of life
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Calisthenic exercise (Experimental): The patients in the calisthenic exercise group will be given one-to-one hands-on calisthenic exercises by the research physiotherapist. They will be asked to do these exercises 3 times a week for 8 weeks. Patients will be followed up by asking whether they do their exercises or not. They will be asked to do the exercises twice a month for 8 weeks under the control of a physiotherapist. In this way, it will be ensured that the exercises are done correctly and that the patients do it completely.
  Interventions: Other: Calisthenic exercise
- Control (No Intervention): Control

INTERVENTIONS:
Other: Calisthenic exercise — Exercises involving major muscle groups will be given. Before starting the calisthenic exercises, they will be asked to perform 10 repetitive warm-ups and breathing exercises. The intensity of the calisthenic exercises will be adjusted on a weekly basis.
  Calisthenic exercises are repeated 10-15 times in the first and second weeks; third and fourth weeks 15-20 repetitive; In the five, six, seven and eight weeks, it will be done with 25-30 repetitions.
  Patients will be asked to keep an exercise diary and weekly follow-ups will be made over the phone.
  Within eight weeks, each patient will come for control twice a month and will be asked to perform the exercises individually under the supervision of a physiotherapist. Patients will be asked to do the exercises three times a week for 8 weeks.
  Arms: Calisthenic exercise

SUMMARY:
The aimed this study is to examine the effects of calisthenic exercises on aerobic capacities, muscle strength and quality of life in patients receiving hemodialysis treatment.

DETAILED DESCRIPTION:
The study is a randomized single-blind placebo-controlled study. . At the beginning and end of the study, all patients will be asked to answer questions including demographic information and a quality of life questionnaire for kidney patients. A 6-minute walking test and a 30-second sit-stand test will be applied by the research physiotherapist to measure their aerobic capacity. Again, a dynamometer will be used to measure muscle strength.

The hypotheses the investigators will test for this purpors; H0 Calisthenic exercise in hemodialysis patients increases aerobic capacity. H1Calisthenic exercise in hemodialysis patients increases muscle strength.H2 Calisthenic exercise in hemodialysis patients improves the quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Being treated in the Hemodialysis unit of Aydın Adnan Menderes University Faculty of Medicine Research and Application Hospital,
* Having good cognitive functions
* Not having regular exercise habits
* Not having a physical disability
* Being between 18-60 years old
* Speaking and understanding Turkish
* Being willing to participate in the study

Exclusion Criteria:

* Neurologically affected patients (such as cerebrovascular accident, Gullian Barre)
* Patients with musculoskeletal problems that prevent exercise
* Patients with advanced heart failure, patients with unstable angina pectoris
* Patients with chronic liver failure
* Patients with a history of cardiovascular events (recent within 12 months)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2023-04-15 (Actual); Study Completion 2023-04-15 (Actual)

PRIMARY OUTCOMES:
Demographic Information Form | immediately after application
  In the form prepared by the researchers with the support of the literature, there are questions about the socio-demographic characteristics of the participants such as gender, age, height, weight, educational status, how long they have been on dialysis, etc.
6 Min. Walking Test | immediately after application
  It is a test method used for the Evaluation of Cardiovascular Endurance. The 6 Minute Walk Test (6MWT) is among the field tests among the cardiopulmonary exercise tests. The test has been proven to be safe, inexpensive and easy to apply. The six-minute walk test is a test that aims to evaluate the submaximal functional capacity by measuring the distance that patients can walk quickly on a hard flat surface in a 6-minute period, in a corridor varying between 30 m and 50 m in length. The 6 MWT is a submaximal exercise test, but correlates well with the maximal cardiovascular exercise test and is better tolerated than other walking tests and better reflects activities of daily living.
30 sec Sit and Stand Test | immediately after application
  30-second sit-stand test to evaluate the dynamic balance and physical fitness lower extremity neuromuscular function levels of individuals It is applied. The test is started while the individual sits in an armless chair, approximately 43 cm high from the ground, in an upright position, with the feet in contact with the ground, with the arms crossed in front of the chest. After the start command is given to the individual, they are asked to come to the standing upright position and again to the sitting position from the determined position for 30 seconds. The number of complete take-offs completed by the individual for 30 seconds is determined.
Grip Force Measurement with Hand Held Dynamometer | immediately after application
  The Jamar Dynamometer is the best known of such devices. During measurements, the hand is in the claw grip position, except for flexion at the metacarpophalangeal joints. The handle part can be adjusted to 5 different levels according to the size of the hand. The Jamar Dynamometer is the most widely used and most reliable grip strength measuring instrument.
Kidney Disease Quality of Life Questionnaire | immediately after application
  This scale is a scale that is used to monitor patients with end-stage rtreatment effects and well-being by self-declaring. assesses quality of life on 8 generics (physical function, role limitations due to social problems, bodily pain, general health, social function, role limitations due to physical problems, energy and fatigue, mental health) and 12 disease-specifi c subscales (effects of kidney disease, symptom list, work status, burden of kidney disease, cognitive function, sexual function, quality of life social interaction, sleep, social support, dialysis staff encouragement, overall health, patient satisfaction). Each subscale is scored out of 100, with higher score indicating greater perceived health al diseasene and evaluates various

CONTACTS AND LOCATIONS:
Overall Officials: Nazan Ozturk, PhD., Principal Investigator — Aydin Adnan Menderes University
Locations (1):
- Aydın Adnan Menderes University Hospital, Aydin, Turkey (Türkiye)